CLINICAL TRIAL: NCT04481932
Title: Trastuzumab Combined With Pyrotinib and Chemotherapy for Locally Advanced, Inflammatory, or Early HER2-positive Mammary glandsCancer: One Arm, Open, Phase II Clinical Study
Brief Title: Trastuzumab Combined With Pyrrolidine and Chemotherapy for Locally HER2 Positive Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, Chairman of Breast Center of Peking University Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-024
Record Dates: First submitted 2020-07-13; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pyrotinib; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab combined with Pyrotinib and chemotherapy (Experimental): The dosage of the above drugs can be adjusted according to the adverse reactions of the subjects. The subject continued to use the drug until the full cycle or the disease progressed or the toxicity was intolerable or withdrawn, or the researcher judged that the medication must be terminated.
  Interventions: Drug: Trastuzumab combined with Pyrotinib and chemotherapy

INTERVENTIONS:
Drug: Trastuzumab combined with Pyrotinib and chemotherapy — Pyrotinib is a small molecule, irreversible tyrosine kinase inhibitor with targets of epidermal growth factor receptor 1 (EGFR/HER1/ErbB1), human epidermal factor receptor 2 (HER2/ErbB2/Neu) and human epidermis Factor Receptor 4 (HER4/ErbB4).
  As a new generation of anti-HER2 therapeutic targeted drugs, pirotinib covalently binds to the ATP binding sites of the kinase regions of EGFR, HER2 and HER4 in cells to prevent homogeneity and heterogeneity of EGFR, HER2 and HER4 in tumor cells Dimer formation, inhibiting its own phosphorylation, blocking the activation of downstream signaling pathways, thereby inhibiting tumor cell growth

SUMMARY:
This study is a one-arm, open, phase II clinical study, and the study subjects are locally advanced and inflammatoryPatients with sexual or early HER2-positive breast cancer entered the trial period after signing informed consentTo evaluate trastuzumab combined with pyrrolitinib and chemotherapy regimen (TCbH+Py) for HER2 positive breastPathologic complete response rate (pCR) for adenocarcinoma.

DETAILED DESCRIPTION:
This study is a single-arm, open, phase II clinical study. The subjects are patients with locally advanced, inflammatory, or early HER2-positive breast cancer. The patients enter the trial period after signing informed consent. This study aims to evaluate trastuzumab The pathological complete response rate (pCR) of anti-combined pyrrotinib and chemotherapy (TCbH+Py) in the treatment of HER2-positive breast cancer.

The subjects began to take continuous medication after joining the group, and the total duration of medication was 6 cycles. Three to four weeks after the end of treatment, the surgeon will choose radical mastectomy, modified radical mastectomy or breast-sparing surgery according to the individual conditions of the patient. Regardless of whether the pCR is achieved, the adjuvant trastuzumab therapy or trastuzumab plus pertuzumab therapy is continued after the operation, and the total course of anti-HER2 therapy is up to 1 year (about 18 treatment cycles). According to the clinical stage and molecular classification of the tumor, it is necessary to decide whether adjuvant radiotherapy, chemotherapy and endocrine therapy are needed.

After the subject finishes all treatments, the subjects who are out of the group for non-PD and non-death causes need to receive the validity Follow-up until PD, start receiving other anti-tumor drug treatment or death (whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

1. Female between 18 and 70 years old;
2. Histologically confirmed as invasive breast cancer;
3. ECOG PS 0-1;
4. The expected survival time is not less than 12 weeks;
5. Standard immunohistochemical HER2-positive breast cancer patients (IHC +++ or FISH amplification);
6. The status of hormone receptors (ER and PR) can be known.
7. Clinical examination or imaging examination of primary lesion >2cm;
8. Patients who are operable (T2-3, N0-1, M0), locally advanced (T2-3,N2-3, M0 or T4A-C, any N, M0) or inflammatory breast cancer (T4d, any N, M0) and who have not received any previous anti-tumor therapy (including radiotherapy, chemotherapy, targeted therapy, except those who have received bisphosphonate therapy previously);
9. Echocardiography indicated left ventricular ejection fraction (LVEF)≥55%;
10. Adequate organ and bone marrow function, as defined below: a. Neutrophil count (ANC)≥ 1,500/mm3 (1.5 × 109/L); B. Platelet count (PLT)≥ 100,000/mm3(100 × 109/L); C. Hemoglobin (Hb)≥ 9 g/dL(90 g/L); D. Serum creatinine ≤ 1.5 times upper limit of normal value (ULN) or creatinine clearance ≥ 60 ml/min(based on Cockroft - Gault formula); E. Total bilirubin (BIL)≤ 1.5 times the upper limit of normal value (ULN); F. AST/SGOT or ALT/SGPT ≤ 2.5 times upper limit of normal value (ULN);G. Urinary protein <2+; If urinary protein ≥2+, 24-hour urinary protein quantification shows protein must1 g or less;
11. I have agreed and signed the informed consent, and am willing and able to comply with the planned visit, research treatment, laboratory examination and other test procedures.

Exclusion Criteria:

1. Have received any previous anti-tumor treatment for primary invasive breast cancer;
2. Previous (<10 years) or other malignant tumors, except for curable cancer species: a. basal cell carcinoma of skin and squamous cell carcinoma b. Carcinoma in situ of cervix
3. For patients with other malignancies, they can also be included in the study if the time from diagnosis to enrollment exceeds 10 years; Prior surgical treatment is permitted except for radiotherapy or systemic therapy (chemotherapy or endocrine therapy);
4. Metastatic breast cancer (M1), bilateral or ipsilateral multifocal breast cancer;
5. Uncontrolled hypertension, systolic blood pressure > 150 MMHG and/or diastolic blood pressure > 100 MMHG), or clinical symptomatic cardiovascular disease, myocardial ischemia and myocardial infarction, severe/unstable angina, poor control of cardiac arrhythmias (including women according to Bazett formula correction QTc interphase < 470 ms), symptoms of congestive heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic cerebral embolism), NYHA Ⅱ magnitude cardiac insufficiency;
6. Receive other anti-tumor treatments within 4 weeks before enrollment;
7. Inability to swallow, intestinal obstruction or other factors affecting the use and absorption of medication;
8. Persons with allergic constitution or known history of allergy to the drug components of the program;
9. The patient has a severe concomitant disease or other conditions that the researcher considers inappropriate for the patient to participate in the studyIn any case;
10. Non-surgically sterilized female patients of childbearing age must have negative serum or urine HCG tests within 14 days prior to study inclusion; And must be non-lactation
11. Other circumstances deemed inappropriate for inclusion by the researcher.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | From enrollment to 18 weeks
  Breast without invasive carcinoma and carcinoma in situ or only carcinoma in situ (ypT0 or ypT0/is)

SECONDARY OUTCOMES:
overall survival (OS) | At least two years
  From the date of enrollment to the time of death due to any cause
Safety index | At least two years
  ECOG PS score, vital signs, physical examination, laboratory examination indicators, ECG, echocardiography, adverse events (AE) according to NCI-CTC AE 5.0 standard

CONTACTS AND LOCATIONS:
Overall Officials: Tao Ouyang, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No